CLINICAL TRIAL: NCT04324307
Title: Multicenter, Open-label Clinical Study of PD-L1/CTLA4 BsAb Combined With Chemotherapy in Locally Advanced and Metastatic Pancreatic Cancer
Brief Title: Study of Immunotherapy Combined With Chemotherapy in Locally Advanced and Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, professor, Changhai Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiH-PP05
Record Dates: First submitted 2020-01-25; First posted 2020-03-27 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced and Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; folfirinox; Oxaliplatin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD-L1/CTLA4 BsAb (Experimental): For 2nd line treatment，PD-L1/CTLA4 BsAb 5mg/kg Q2W
  Interventions: Drug: PD-L1/CTLA4 BsAb
- PD-L1/CTLA4 BsAb + GP (Experimental): For 1st line treatment，PD-L1/CTLA4 BsAb 5mg/kg Q2W in combination with Gemcitabine 1000 mg/m2 and Nab-paclitaxel 125 mg/m2 , 28days/cycle
  Interventions: Drug: PD-L1/CTLA4 BsAb; Combination Product: GP
- PD-L1/CTLA4 BsAb + FOLFIRINOX (Experimental): For 1st line treatment，PD-L1/CTLA4 BsAb 5mg/kg Q2W in combination with Oxaliplatin 68 or 85 mg/m2, Irinotecan 135 or 150 or 180 mg/m2, Calcium Folate 400 mg/m2, Fluorouracil 2400mg/m2, 14 days/cycle
  Interventions: Drug: PD-L1/CTLA4 BsAb; Combination Product: FOLFIRINOX

INTERVENTIONS:
Drug: PD-L1/CTLA4 BsAb — PD-L1/CTLA4 BsAb 5mg/kg, iv，Q2W
Combination Product: GP — Gemcitabine 1000mg/m2, iv, D1,8,15, 28days/cycle; nab-Paclitaxel 125mg/m2，iv，D1,8,15, 28days/cycle;
  Other Names: Gemcitabine; nab-Paclitaxel
  Arms: PD-L1/CTLA4 BsAb + GP
Combination Product: FOLFIRINOX — Fluorouracil 2400mg/m2，iv，D1, 14days/cycle; Oxaliplatin 68-85mg/m2，iv, D1,14days/cycle;Irinotecan135-180mg/m2，iv, D1, 14days/cycle;Calcium Folate 400mg/m2，iv, D1, 14days/cycle;
  Other Names: Oxaliplatin; Irinotecan; Calcium Folate; Fluorouracil
  Arms: PD-L1/CTLA4 BsAb + FOLFIRINOX

SUMMARY:
To evaluate the efficacy of PD-L1/CTLA4 BsAb for the second line treatment and the combination with chemotherapy for the first line treatment in pancreatic cancer

DETAILED DESCRIPTION:
Subjects who signed the informed consent were assigned to three cohorts according to the actual treatment status. Cohort 1 enrolled subjects receiving PD-L1/CTLA4 BsAb 5mg/kg iv Q2W for 2nd treatment; cohort 2 enrolled subjects receiving PD-L1/CTLA4 BsAb in combination with gemcitabine/albumin- paclitaxel as 1st treatment for 4-6 cycles with PD-L1/CTLA4 BsAb monotherapy maintainence; cohort 3 enrolled subjects received systemic chemotherapy, receiving PD-L1/CTLA4 BsAb combined with oxaliplatin / irinotecan / leucovorin / fluorouracil (FOLFIRINOX) as 1st treatment for 4-6 cycles withPD-L1/CTLA4 BsAb monotherapy maintainence; until disease progression according to RECIST 1.1, intolerable toxicity, withdrawal, death, 2-yr treatment,who comes first.

ELIGIBILITY:
Inclusion Criteria:

* Histology or cytology confirmed as pancreatic ductal adenocarcinoma;
* ECOG 0-1;
* adequate organ function (absolute neutrophil count ≥1.5 x 109/L; platelet count ≥100 x 109/L; creatinine < 1.5 x ULN (upper normal) or calculated creatinine clearance ( CRCI) ≥ 60mL/min; albumin ≥ 30g/L; total bilirubin <1.5 x ULN; aspartate aminotransferase (AST) < 2.5 x ULN; alanine aminotransferase (ALT) < 2.5x ULN; INR or PT < 1.5x ULN, and aPTT <1.5x ULN);
* no obvious symptoms of jaundice and ascites;
* no other serious underlying diseases

Exclusion Criteria:

* patients with active brain metastases;
* history of autoimmune diseases, or need to be treated with corticosteroids and immunosuppressive agents;
* past history of unstable angina, symptomatic congestive heart failure, severe arrhythmia, myocardial infarction within 6 months, QT interval prolongation (>450ms);
* other malignant tumors within the last 5 years;
* pregnant or lactating women;
* NRS ≥ 4 points;
* unintentional weight loss ≥ 5% within 1 month before the first dose even if peripheral or central vein nutrition support,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  objective response rate

SECONDARY OUTCOMES:
DCR | 2 years
  Disease Control Rate
DOR | 2 years
  Duration of Response
TTP | 2 years
  Time to Response
PFS | 2 years
  Progression Free Survival
OS | 2 years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, Doctor, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China